CLINICAL TRIAL: NCT05554874
Title: Effect of Pulsed Electromagnetic Stimulation on DOMS: A Randomized Sham-controlled Trial.
Brief Title: Effect of Pulsed Electromagnetic Stimulation on DOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Nur OYMAK SOYSAL, Principal investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.05.2022/08
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Electromagnetic Fields
Keywords: Electromagnetic Fields; Delayed Onset muscle soreness

STUDY DESIGN:
Intervention Model Description: Real or sham pulsed electromagnetic fields
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): participants undergoing pulsed electromagnetic fields
  Interventions: Other: Pulsed electromagnetic fields
- Control group (Sham Comparator): participants undergoing sham pulsed electromagnetic fields
  Interventions: Other: Sham Pulsed electromagnetic fields

INTERVENTIONS:
Other: Pulsed electromagnetic fields — receiving Pulsed electromagnetic fields 3 times, immediately after the onset of delayed muscle soreness, 24 and 48 hours later.
  Arms: Case group
Other: Sham Pulsed electromagnetic fields — Sham application will be applied with the same device without applying magnetic current.
  Arms: Control group

SUMMARY:
The aim of our study is to investigate the effect of Pulsed Electro Magnetic Field application on delayed muscle soreness in healthy Quadriceps femoris muscle.

DETAILED DESCRIPTION:
Participants will complete 100 consecutive fall jumps from a 0.60 m high platform to generate Delayed muscle soreness. After landing, participants will be encouraged to jump vertically immediately with maximum force. Five sets of 20 jumps will be performed with 10-second intervals between each jump, with a 2-minute rest between sets.Immediately after the implementation of the exercise protocol that will cause delayed muscle soreness, the participants will be randomly divided into 2 groups. Pulsed Electromagnetic Field or sham Pulsed Electromagnetic Field application will be applied to the non-dominant extremities of the participants.

The participants will be evaluated before (0), 24, 48 and 72 hours after the delayed muscle pain protocol.

Pain intensity of the participants will be evaluated with Visual Pain Scale (VAS), muscle fatigue will be evaluated with Modified Borg Scale, muscle performance will be evaluated with one-leg jump test, and muscle tenderness will be evaluated with an algometer.

In addition, serum creatine kinase and myoglabin values will be tested by laboratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* not having any systemic disease
* not having neuromuscular deficit
* not having knee pathology
* To be defined as inactive (less than 30 minutes of moderate physical activity five times a week) according to the minimum activity guidelines published by the American College of Sports Medicine

Exclusion Criteria:

* Being actively involved in any sport
* participating in a regular exercise program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Pain intensty | up to 72 hours
  assessed with VAS
Muscle fatigue | up to 72 hours
  Borg scale
Muscle performance | up to 72 hours
  Single leg hop test
Muscle tenderness | up to 72 hours
  Algometer

CONTACTS AND LOCATIONS:
Overall Officials: Ummuhan Bas Aslan, Prof, Study Chair — Prof Dr.
Locations (1):
- Ayşe Nur Oymak Soysal, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nosaka K, Newton M, Sacco P. Delayed-onset muscle soreness does not reflect the magnitude of eccentric exercise-induced muscle damage. Scand J Med Sci Sports. 2002 Dec;12(6):337-46. doi: 10.1034/j.1600-0838.2002.10178.x. PMID 12453160
- [Background] Sellwood KL, Brukner P, Williams D, Nicol A, Hinman R. Ice-water immersion and delayed-onset muscle soreness: a randomised controlled trial. Br J Sports Med. 2007 Jun;41(6):392-7. doi: 10.1136/bjsm.2006.033985. Epub 2007 Jan 29. PMID 17261562
- [Background] 11. Rasmussen, C., Rathleff, M. S., Knudsen, C., Skou, S. T., Jørgensen, M., Olesen, J., et al. (2012). Pulsed electromagnetic field therapy reduces delayed onset muscle soreness in marathon runners. In A double-blind randomized placebo-controlled study. 13th EFORT (pp. 1e18).
- [Background] 12. Walsh, J., Simonds, L., & Tiidus, P. (2010). Pulsed magnetic field therapy does not influence indices of muscle damage following eccentric exercise: a preliminary study. Medicine in Sport, 14(4), 199e203.